CLINICAL TRIAL: NCT04318340
Title: A Novel Tapered Applicator for Post-Hysterectomy Vaginal Vault Brachytherapy: Quality-of-Life Assessment of Patient Comfort and In Vivo Dosimetry
Brief Title: A Novel Tapered Applicator for Vaginal Vault Brachytherapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 2000026385
Record Dates: First submitted 2020-03-20; First posted 2020-03-23 (Actual); Last update posted 2023-07-14 (Actual); Status verified 2023-07

CONDITIONS: Endometrial Cancer; Brachytherapy; Quality of Life
MeSH Terms: conditions — Endometrial Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Applicators (Active Comparator): All patients will be fitted with the 2.6 cm applicator and sized up to the 3.0 cm applicator if tolerable.
  Interventions: Other: Standard applicator
- Tapered Applicator (Experimental): All patients will be fitted with the novel tapered 3.0 cm applicator. Patients have the option of having magnetic resonance imaging with the tapered applicator in place.
  Interventions: Other: Tapered applicator

INTERVENTIONS:
Other: Tapered applicator — An applicator inserted in 2 steps that tapers at the distal vagina
  Arms: Tapered Applicator
Other: Standard applicator — A 2.6 cm standard applicator is inserted and sized up to a standard 3 cm applicator if tolerable.
  Arms: Standard Applicators

SUMMARY:
This study will assess the comfort and fit of a novel applicator for endometrial cancer patients who are candidates for vaginal brachytherapy. This study is only assessing the applicator fitting. No patients in this study will be treated with the novel applicator.

DETAILED DESCRIPTION:
In the treatment of endometrial cancer, adjuvant vaginal brachytherapy is typically performed to deliver radiation dose to the apex of the vagina with a fixed diameter vaginal applicator which extends the full length of the vagina. The largest cylinder which fits at the apex provides the best dosimetry. Smaller diameter cylinders may provide sub-optimal coverage of potential areas of disease. Due to pain or discomfort with a large cylinder, some women may be treated with a smaller diameter cylinder. A novel applicator, with a tapered design and two-step insertion was fabricated to improve the comfort, fit, and patient compliance of this procedure while maintaining optimum geometry and dosimetry at the dome. Our primary aim is to assess patient comfort with the new applicator. Patients will be fit with different applicators (standard of care and novel tapered vaginal applicator) and their comfort will be assessed with a visual analog scale-based survey, comparing the two.

Aim #1: Assess if the 3.0cm diameter novel tapered applicator is more comfortable than the standard 3.0cm diameter applicator among patients fitted with a standard 3.0cm diameter applicator.

Aim #2: Determine what percentage of patients who would otherwise be treated with a standard 2.6cm diameter vaginal cylinder can be up-sized to a 3.0cm diameter cylinder with the novel tapered applicator design.

Aim #3: Assess in vivo dosimetry (optional for all patients). Patients who are prescribed vaginal brachytherapy undergo 3-dimensional cross-sectional imaging (i.e., MRI or CT) prior to treatment, as standard of care. This is done with the standard treatment applicator inserted to assess radiation dose distribution. In this optional aim, patients will undergo a slightly longer MRI, with additional MRI images performed with the novel tapered applicator in place to characterize and assess dosimetry, fit, contact with mucosal surfaces and presence of air gaps in comparison to a standard cylindrical applicator.

ELIGIBILITY:
Eligibility Criteria

* Patients with stage I-IV endometrial cancer.
* Patient must have been treated with hysterectomy.
* A radiation oncology determined the patient's disease warrants adjuvant treatment with vaginal brachytherapy as sole adjuvant radiotherapy.
* Patient consented to receive standard of care vaginal brachytherapy treatment.
* Vaginal cuff deemed healing appropriately by treating radiation oncologist during initial consultation without evidence of infection, pelvic symptoms, or other surgical complications.
* 18 ≤ Age
* English speaking.

Exclusion Criteria

* Subjects meeting any of the criteria below may not participate in the study:
* Requires premedication with pain medications and/or anxiolytics during applicator fitting.
* Will receive pelvic EBRT.
* Prior known diagnosis of lupus, scleroderma, dermatomyositis, Crohn's disease, ulcerative colitis, pacemakers, or other contraindications to radiotherapy.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2020-07-16 (Actual); Primary Completion 2023-03-20 (Actual); Study Completion 2023-03-20 (Actual)

PRIMARY OUTCOMES:
Patient comfort | up to 10 minutes
  Patient comfort will be assessed with a visual analog scale-based survey rating 0 (none) to 10 (severe) in each of the following domains: pain, pressure, burning, stress, hardness/roughness, and stretching at both insertion and in final resting positions.
Ability to up-size with tapered applicator | up to 10 minutes
  Determine what percentage of patients who would otherwise be treated with a standard 2.6cm diameter vaginal cylinder can be up-sized to a 3.0cm diameter cylinder with the novel tapered applicator design.

SECONDARY OUTCOMES:
Assess in vivo dosimetry (optional for all patients) | up to 10 minutes
  Patients who are prescribed vaginal brachytherapy undergo 3-dimensional cross-sectional imaging (i.e., MRI or CT) prior to treatment, as standard of care. This is done with the standard treatment applicator inserted to assess radiation dose distribution. In this optional aim, patients will undergo a slightly longer MRI, with additional MRI images performed with the novel tapered applicator in place to characterize and assess dosimetry, fit, contact with mucosal surfaces and presence of air gaps in comparison to a standard cylindrical applicator.

CONTACTS AND LOCATIONS:
Overall Officials: Shari Damast, MD, Principal Investigator — Yale University
Locations (1):
- Smilow Cancer Hospital, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No